CLINICAL TRIAL: NCT00005489
Title: Salt Sensitivity, Cardiovascular and Metabolic Disease
Status: Completed | Type: Observational
Sponsor: Indiana University (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Other Study IDs: 5005; R01HL057826 (NIH)
Record Dates: First submitted 2000-05-25; First posted 2000-05-26 (Estimated); Last update posted 2015-12-30 (Estimated); Status verified 2015-12

CONDITIONS: Cardiovascular Diseases; Heart Diseases; Hypertension; Angina Pectoris; Cerebrovascular Accident; Myocardial Infarction; Diabetes Mellitus; Heart Failure, Congestive; Heart Failure
MeSH Terms: conditions — Cardiovascular Diseases; Heart Diseases; Hypertension; Angina Pectoris; Stroke; Myocardial Infarction; Diabetes Mellitus; Heart Failure

SUMMARY:
To identify the role of salt-sensitivity of blood pressure in the pathogenesis of hypertension.

DETAILED DESCRIPTION:
DESIGN NARRATIVE:

Approximately 498 of 750 normal and hypertensive subjects who were carefully characterized in terms of blood pressure response to salt loading and depletion in the late 1970s were re-examined to identify physiological factors contributing to salt-sensitivity of blood pressure. This helped to confirm preliminary observations suggesting that salt sensitivity in normotensive subjects predicted the subsequent development of hypertension with aging. In addition, longitudinal observations in hypertensive patients and in normotensives helped to determine whether salt-sensitivity or salt-resistance of blood pressure were associated with differences in the risk for development of specific forms of cardiovascular disease (stroke, angina, myocardial infarction, congestive heart failure), renal and metabolic (diabetes mellitus) disorders.

ELIGIBILITY:
No eligibility criteria

Max Age: 100 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 1998-01; Study Completion 2001-12

CONTACTS AND LOCATIONS:
Overall Officials: Myron Weinberger — Indiana University-Purdue University

REFERENCES:
- [Background] Weinberger MH, Fineberg NS, Fineberg SE, Weinberger M. Salt sensitivity, pulse pressure, and death in normal and hypertensive humans. Hypertension. 2001 Feb;37(2 Pt 2):429-32. doi: 10.1161/01.hyp.37.2.429. PMID 11230313
- [Background] Weinberger M, Weinberger MH, Fineberg N, Fineberg SE, Wagner U. Long-term follow-up of participants in clinical studies. J Clin Epidemiol. 2002 Mar;55(3):230-4. doi: 10.1016/s0895-4356(01)00437-1. PMID 11864792
- [Background] Weinberger MH, Fineberg NS, Fineberg SE. The influence of blood pressure and carbohydrate tolerance on vascular compliance in humans. Am J Hypertens. 2002 Aug;15(8):678-82. doi: 10.1016/s0895-7061(02)02955-2. PMID 12160189
- [Background] Weinberger MH. Salt sensitivity is associated with an increased mortality in both normal and hypertensive humans. J Clin Hypertens (Greenwich). 2002 Jul-Aug;4(4):274-6. doi: 10.1111/j.1524-6175.2002.00924.x. PMID 12147930
- [Background] Weinberger MH, Fineberg NS, Fineberg SE. Effects of age, race, gender, blood pressure, and estrogen on arterial compliance. Am J Hypertens. 2002 Apr;15(4 Pt 1):358-63. doi: 10.1016/s0895-7061(02)02261-6. PMID 11991223